CLINICAL TRIAL: NCT07031765
Title: Peds CHAMP1ON - Combinatorial Hematopoietic Stem Cell And Monoclonal Antibody PD-1 Blockade Phase 1 Trial for RecurreNt Pediatric High-Grade Glioma
Brief Title: Peds CHAMP1ON - Hematopoietic Stem Cell And Monoclonal Antibody PD-1 Blockade for RecurreNt Pediatric High-Grade Glioma
Acronym: Peds CHAMP1ON
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20252524; OCR47280 (Other: University of Florida)
Record Dates: First submitted 2025-06-02; First posted 2025-06-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Recurrent High-grade Glioma; Grade III Astrocytoma; Oligodendroglioma; Oligoastrocytoma; Ependymoma; Grade IV Astrocytoma
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Ependymoma; Glioblastoma | interventions — Nivolumab; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adjuvant exHSCs + Nivolumab (starting after surgery/biopsy) (Arm 1) (Experimental): Immediate maximal surgical resection or biopsy, untreated tumor. exHSCs and Nivolumab will be administered after maximal surgical resection.
  Interventions: Biological: exHSC; Drug: Nivolumab; Procedure: Resection or biopsy
- Neoadjuvant exHSCs + Nivolumab (starting before surgery/biopsy) (Arm 2) (Experimental): exHSCs + Nivolumab will be administered prior to maximal surgical resection or biopsy.
  Interventions: Biological: exHSC; Drug: Nivolumab; Procedure: Resection or biopsy

INTERVENTIONS:
Biological: exHSC — Ex vivo expanded CD34+ hematopoietic stem cells (exHSCs) at a targeted dose of 2.5 x 106 cells/kg (or maximal achievable dose, with a minimum deliverable dose of 1/10 target dose; max dose 1.0 x 108 total cells for patients ≥40kg).
Drug: Nivolumab — Nivolumab 3mg/kg once every 2 weeks, max dose 240mg. Nivolumab will be administered on day 1 and day 15 of each cycle for a total of 10 cycles. Nivolumab may continue for a total two years of therapy, at the discretion of the treating team.
Procedure: Resection or biopsy — Patients must be candidates for standard of care surgical resection or biopsy.

SUMMARY:
This is a Phase I study of ex vivo expanded CD34+ hematopoietic stem cells (exHSCs) plus nivolumab in pediatric patients with histologically confirmed diagnosis of a non-brainstem high-grade glioma (NB-HGG, WHO Grade III or IV astrocytoma, oligodendrogliomas, oligoastrocytomas, ependymomas) that is recurrent, progressive or refractory following radiotherapy with or without chemotherapy. Patients must be candidates for standard of care surgical resection or biopsy.

DETAILED DESCRIPTION:
This is a Phase I study of ex vivo expanded CD34+ hematopoietic stem cells (exHSCs) plus nivolumab in pediatric patients with recurrent high-grade glioma. One cycle will be 28 days in length with exHSCs + Nivolumab being administered on day 1 and Nivolumab alone being administered on day 15 of each cycle for a total of 10 cycles. Nivolumab may continue for a total two years of therapy, at the discretion of the treating team.

There are two arms: Arm 1 - Immediate maximal surgical resection or biopsy, untreated tumor. exHSCs and Nivolumab will be administered after maximal surgical resection. Arm 2 - exHSCs + Nivolumab will be administered prior to maximal surgical resection or biopsy. exHSCs + Nivolumab will be administered after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of a non-brainstem high-grade glioma (NB-HGG, WHO Grade III or IV astrocytoma, oligodendrogliomas, oligoastrocytomas, ependymomas) that is recurrent, progressive or refractory following radiotherapy with or without chemotherapy. Patients must be candidates for standard of care surgical resection or biopsy.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in two dimensions.
* Patients must have recovered from the acute treatment related toxicities (defined as ≤ grade 2 if not defined in eligibility criteria) of all prior chemotherapy, immunotherapy, radiotherapy or any other treatment modality prior to entering this study.
* Patients must have received their last dose of known myelosuppressive anticancer therapy greater than 21 days prior to enrollment.
* Patients must have received their last dose of the investigational or biologic agent ≥ 7 days prior to study enrollment.

  * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration must be discussed with and approved by the study chair.
  * Monoclonal antibody treatment and/or agents with prolonged half-lives: At least three half-lives must have elapsed prior to enrollment.
* Patients must have had their last fraction of:

  * Craniospinal irradiation ≥ 3 months prior to enrollment.
  * Other substantial bone marrow irradiation ≥6 weeks prior to enrollment
  * Local palliative XRT ≥2 weeks
* ≥ 12 weeks since autologous bone marrow/stem cell transplant prior to enrollment

  *Patients with any history of allogeneic transplant are not eligible
* Patient must be ≥ 4 but ≤ 26 years of age at the time of enrollment.
* Karnofsky ≥ 60% for > 16 years of age; Lansky ≥ 60% for children ≤ 16 years of age

  • Participants who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Patients must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count >1000 cells/μL
  * Platelets >75,000 cells/μL(unsupported, defined as no platelet transfusion within 7 days)
  * Hemoglobin ≥8g/dl (may receive transfusions)
  * Total bilirubin ≤1.5 times institutional upper limit of normal (ULN)
  * ALT(SGPT) <3 x institutional upper limit of normal
  * Albumin ≥2 g/dl
  * Serum creatinine based on age/gender as noted in Table 1 Patients that do not meet the criteria below but have a 24hour Creatinine Clearance or GFR (radioisotope or iothalamate) ≥ 70 ml/min/1.73 m2 are eligible.
  * INR or PT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Pulmonary function - Pulse oximetry > 93% on room air and no evidence of dyspnea at rest.
* Patient must be a candidate for surgical resection or biopsy at the time of enrollment. The goal of surgical resection is both cytoreduction and tumor debulking, or biopsy for diagnosis confirmation as part of standard of care.
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to enrollment. A baseline detailed neurological exam should clearly document the neurological status of the patient at the time of enrollment on the study.
* Patients must be on a stable or decreasing dose of corticosteroids for 7 days prior to enrollment. A maximum dexamethasone dose of 0.1 mg/kg/day is allowed (4 mg maximum), but preferably have been discontinued (inhaled or topical use of steroids is allowed).
* The effects of nivolumab on the developing human fetus are unknown. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months after completion of nivolumab administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 5 months after completion of nivolumab administration.

Female subjects of childbearing potential must not be pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

- Ability to understand and the willingness to sign a written informed consent document. Parents/Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Patients with evidence of leptomeningeal, primary spinal cord, or multicentric disease.
* Patients who have not recovered to ≤ Grade 1 or baseline from adverse events due to prior anti-cancer therapy.
* Patients who are receiving any other investigational agents.
* Female subjects of childbearing potential must not be pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab.
* Prior treatment with an anti-PD-1, anti PD-L1 and anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Patients who have had prior allogenic hematopoietic stem cell transplant.
* Participants with an active, known, or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Patients with uncontrolled intercurrent illness or any other significant condition(s) (serious infections or significant psychiatric, cardiac, pulmonary, hepatic, or other organ dysfunction that in the opinion of the investigator would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity, or would interfere with the study procedures or results.
* Patients who have had live vaccines within 30 days prior to the first dose of trial treatment.

Ages: 4 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Rate of DLTs in treated participants | At the end of Cycle 1 (each cycle is 28 days)
  Rate of DLTs in participants treated with exHSCs + αPD-1. Cycle 1 Day 1 is the first day exHSCs + Nivo is given.
Rate of ability to manufacture a product that meets release specifications and deliver the first study treatment | At the end of Cycle 1 (each cycle is 28 days)
  Feasibility of delivering exHSCs + αPD-1. Cycle 1 Day 1 is the first day exHSCs + Nivo is given.

CONTACTS AND LOCATIONS:
Overall Officials: John Ligon, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Children's Hospital/Shands Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No